CLINICAL TRIAL: NCT07373106
Title: SHORT-TERM EFFECTS OF BROCCOLI-DERIVED GLUCORAPHANIN ON RECOVERY FROM ECCENTRIC MUSCLE DAMAGE: A DOUBLE-BLIND RANDOMIZED CROSSOVER STUDY
Brief Title: Short-term Effects of Broccoli-derived Glucoraphanin on Recovery From Eccentric Muscle Damage
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian Sports University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MNLKIN(M)-2024-574
Record Dates: First submitted 2025-09-15; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- male volunteers aged 18-35 years (Experimental)
  Interventions: Dietary Supplement: broccoli powder consumption; Dietary Supplement: Placebo (no broccoli-derived bioactives)

INTERVENTIONS:
Dietary Supplement: broccoli powder consumption — Participants underwent two separate sessions of muscle-damaging exercise targeting the elbow flexors: (1) following seven days of broccoli powder consumption (condition X), and (2) following an equivalent placebo regimen (condition Y). The broccoli supplementation consisted of 10 g of broccoli powder [a freeze-dried glucoraphanin-rich broccoli powder (99.5% broccoli and 0.5% mustard seed)] dissolved in 125 mL of boiling water, providing 320 μg of glucoraphanin per serving. It was consumed when still hot/warm once daily for seven days before and for four days following the eccentric exercise protocol. The placebo powder, matched in appearance and preparation, contained no broccoli-derived bioactives.
Dietary Supplement: Placebo (no broccoli-derived bioactives) — The placebo powder, matched in appearance and preparation, contained no broccoli-derived bioactives.

SUMMARY:
Eccentric exercise induces muscle damage and delay functional recovery. Broccoli-derived glucoraphanin (a sulforaphane precursor that activates Nrf2 defenses) may aid repair; however, its short-term effects in humans remains unknown. This study aims to evaluate whether short-term supplementation with broccoli-derived glucoraphanin will improve recovery from exercise-induced muscle damage. In a randomized, double-blind, placebo-controlled crossover design, fifteen participants will consume either high-glucoraphanin broccoli powder (320 μg) or placebo for one week, followed by elbow flexor eccentric exercise and continued supplementation. Strength, soreness, creatine kinase (CK), range of motion (ROM), arm girths, and ultrasound-assessed muscle and tendon morphology will be measured at baseline, immediately post-exercise, and at 48 and 96 hours post-exercise.

ELIGIBILITY:
Inclusion Criteria:

* no resistance training experience in the past 6 months, no arm injuries in the past 2 years, no illnesses in the month prior to data collection, and no known allergies to broccoli or other cruciferous vegetables.

Exclusion Criteria:

* incomplete participation.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Peak torque, Nm/s | At baseline, immediately post-exercise, and at 48 hours, and at 96 hours post-exercise.
  Exercise induced damage marker, isokinetic and isometric knee extension
Range of motion, degree | At baseline, immediately post-exercise, and at 48 hours, and at 96 hours post-exercise.
  Exercise induced damage marker, elbow extension and flexion
Arm girth, mm | At baseline, immediately post-exercise, and at 48 hours, and at 96 hours post-exercise.
  Exercise induced muscle damage marker, arm relaxed and fully flexed

SECONDARY OUTCOMES:
Soreness, points | At baseline, immediately post-exercise, and at 48 hours, and at 96 hours post-exercise.
  exercise induced damage marker, biceps brachii, 10-point visual analogue scale with 0 indicating no soreness and 10 indicating intolerably intense soreness.
Creatine kinase, IU/L | At baseline, immediately post-exercise, and at 48 hours, and at 96 hours post-exercise.
  Exercise induced muscle damage marker in venous blood

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: version 1 (2025-09-15): https://cdn.clinicaltrials.gov/large-docs/06/NCT07373106/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan: version 2 (2025-09-26): https://cdn.clinicaltrials.gov/large-docs/06/NCT07373106/Prot_SAP_001.pdf